CLINICAL TRIAL: NCT04415528
Title: Emotion-Focused Mindfulness Therapy: A Feasibility Study for Late Life Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stacey Hatch (Other)
Responsible Party: Sponsor-Investigator, Stacey Hatch, Stacey Hatch, PhD candidate, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1509
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Anxiety
Keywords: anxiety; aging and health; adults aged 65 and older; mindfulness based intervention; meditation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This will be a small pilot RCT study that will use a wait list control trial design. Participants will be randomly allocated to either the intervention or control group
Who Masked: Outcomes Assessor
Masking Description: This study involves partial disclosure to prevent confirmation bias on the part the research assistant who will be administering assessments. The research assistant will be blinded to the study purpose throughout the study. Participants will be informed that there will be different phases of data collection, and provision of the intervention. The research assistant will not be informed of participant allocation to the intervention group or the wait list control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will begin receiving the group intervention within one - two weeks of Time 1 assessment. This group will receive Time 2 assessments at the end of the group delivery. Time 3 assessments will be administered eight weeks after the completion of group delivery.
  Interventions: Other: Emotion-Focused Mindfulness Therapy
- Wait listed control group (Active Comparator): The wait listed control group will be assessed at Time 1, eight weeks before receiving the intervention. This group will receive Time 2 assessments at the beginning of their group delivery. This group will complete Time 3 assessments eight weeks after the completion of group delivery.
  Interventions: Other: Emotion-Focused Mindfulness Therapy

INTERVENTIONS:
Other: Emotion-Focused Mindfulness Therapy — EFMT is a group intervention of 8weekly meetings of 2.5 hours with 10 - 12 participants per group. Participants are provided instruction that encourages noting and experiencing bodily sensations and emotions during meditations. Meditations are conducted in silence for between 20 and 35 minutes. Participants are asked to journal their recollection of the meditation and experiences that arise for them as they journal. Each participant then describes their experience in meditation, with the facilitator offering empathic exploration to support transforming negative emotions into adaptive emotions.
  The study will be conducted in an online PHIPPA protected platform and has been modified to accommodate electronic delivery. Maximum number of participants per group will be six, and each session will be 1.5 hours. Data will be collected at three points by a research assistant to evaluate the feasibility of EFMT for older adults and determine whether anxiety is influenced by the intervention.

SUMMARY:
Canadians 65 and older experience anxiety at a rate of 6.4%, affecting more than 300,000 people. In Ontario, 5.6% of adults 65 and older have anxiety, representing over 100,000 people. Eastern Ontario primary care clinics report significantly higher numbers of adults 65 and older diagnosed with anxiety at between 28% and 30%, representing approximately 4,600 people diagnosed with anxiety. Costs to the Canadian health care system of anxiety in community dwelling adults aged 65 and older have been estimated at $61.2 to $119.8 million per 1,000,000 people. These costs can reasonably be expected to increase by 2021 when the percentage of older adults 65+ with mental illness is estimated to be approximately 30% of the older population base.

Anxiety in older adults has been linked retaining new information and the instrumental activities of daily living, sleep disturbance, suicidal ideation particularly among men, and increased use of health care services. Present pharmacological treatments for anxiety in older adults have met with limited success. Mindfulness-based interventions (MBIs) are an area of research interest in the treatment of anxiety. The use of MBIs has shown a trend toward self-reported lower levels of chronic stress and psychological stress among older adults small scale RCTs and qualitative studies.

Emotion focused mindfulness meditation therapy (EFMT) is a MBI that shows promise. EFMT has been demonstrated to reduce symptoms of anxiety in general populations. EFMT's focus on meditation and the felt sense of emotions, rather than learning new material, may make it a promising intervention for reducing symptoms of anxiety for older adults who often report normal aging problems such as general forgetfulness and difficulty with word recall. EFMT may be a potentially promising intervention that has not yet been tested in older adults. EFMT can be offered in primary care, community and hospital settings. Further research is required to determine if EFMT could reduce anxiety for older adults.

DETAILED DESCRIPTION:
The purpose of this small scale RCT is to determine the feasibility and acceptability of EFMT among community dwelling older adults who experience anxiety. This study has the following three aims: to determine if participants can be recruited, enrolled, and retained; to determine if participants can adhere to all components of the intervention; and to determine the extent to which participants who receive the intervention have decreased levels of anxiety compared to those who do not receive the intervention. The secondary outcomes will be to determine the extent to which participants who receive the intervention have improved sleep quality, and improved subjective memory functioning compared to those who do not receive the intervention.

This will be a small pilot RCT study that will use a wait list control trial design. Participants will be randomly allocated to either the intervention or control group. Emotion-Focused Mindfulness Therapy (EFMT) is a group intervention consisting of eight weekly meetings of 2.5 hours with 10 - 12 participants per group. Participants are provided instruction that encourages noting and experiencing bodily sensations and emotions during meditations. Meditations are conducted in silence for between twenty and thirty-five minutes, and then participants are asked to journal their recollection of the meditation and experiences that arise for them as they journal. Following journalling, each participant describes their experience in meditation, with the facilitator offering empathic exploration to support transforming negative emotions into adaptive emotions.

The study will be conducted in an online delivery PHIPPA protected platform and has been modified to accommodate electronic delivery. Maximum number of participants per group will be six, and each session will be 1.5 hours. Data will be collected at three points by a research assistant to evaluate the feasibility of EFMT for older adults and determine whether anxiety is influenced by the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be community dwelling older adults at least 65 years of age and with have no existing therapeutic alliance with the PI. Inclusion criteria will be a diagnosis or self-report of anxiety. The presence of symptoms of anxiety will be assessed using the Geriatric Anxiety Inventory (GAI) with a cut off score of 10 which indicates the presence of anxiety (Johnco et al., 2015). Participants will be willing to commit to an eight-week program.

Exclusion Criteria:

* Exclusion criteria will be beginning or stopping psychotropic medications within the previous six weeks and concurrent participation in any other mindfulness-based group during the study. Participants will not be excluded if they have prior experience with mindfulness. Further exclusion criteria will be a Telephone Montreal Cognitive Assessment (T-MoCA) cut off score of 19 which indicates the possibility of mild cognitive impairment.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Determine if participants can be recruited, enrolled, and retained | 8 weeks
  Data will be gathered and measured on the number of potential participants referred and screened for eligibility, participants meeting eligibility requirements, participants enrolled, and participants completing the intervention. Dates defining the recruitment period will be reported. Number of participants referred by physicians and number of participants who call the PI directly will be combined for each site.
Determine if participants can adhere to all components of the intervention | From time of enrollment to end of intervention at 8 weeks
  To determine if participants can adhere to the intervention, attendance of 6 / 8 sessions, data on attendance will be gathered. Data for the other measures of adherence of meditation, journaling and reporting will also be gathered. In the tradition of MBI research, the intervention will be considered complete if participants are able to attend a minimum of six of eight meetings (Santorelli, Florence Meleo-Meyer, Koerbel, & Kabat-Zinn, 2017). Data gathered on adherence to meditation, journaling and reporting aspects of the intervention through weekly reporting forms to be completed by each participant through an online survey. Participants will answer yes or no to whether they engaged in each component. Participants are not required to practice at home, however data will be gathered on the frequency and duration of home practice meditation and journaling to determine if there is a relationship to outcomes.
Geriatric Anxiety Inventory, to assess change over time | Time 1: at enrollment; Time 2: end of intervention at 8 weeks; Time 3: 8 weeks post-intervention
  The Geriatric Anxiety Inventory (GAI) consists of 20 "Agree/Disagree" items designed to assess typical common anxiety symptoms.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PQSI) to to assess change over time | Time 1: at enrollment; Time 2: end of intervention at 8 weeks; Time 3: 8 weeks post-intervention
  The PQSI is a questionnaire validated for use with community dwelling older adults (Carpenter & Andrykowski, 1998). This measure was selected because sleep complaints are frequently associated with anxiety (C.-M. Yang, Lo, & Spielman, 2006).The PQSI is a simple 19 item subjective measure of sleep quality and patterns of sleep using a 0 to 3 Likert scale (Smyth, 2008).
Multifactorial Memory Questionnaire (Troyer & Rich, 2002), to assess change over time | Time 1: at enrollment; Time 2: end of intervention at 8 weeks; Time 3: 8 weeks post-intervention
  The Multifactorial Memory Questionnaire (MMQ) is a self-assessment scale that measures three aspects of metamemory. Items are scored on a 5-point Likert scale (Troyer & Smith, 2018).

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Hatch, PhDcandidate, Principal Investigator — Queens University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gayner, B. (2019). Emotion-focused mindfulness therapy. Person-Centered & Experiential Psychotherapies, 1-23. https://doi.org/10.1080/14779757.2019.1572026
- [Background] Statistics Canada. (2012). Table 13-10-0465-01: Mental health indicators. https://doi.org/https://doi.org/10.25318/1310046501-eng
- [Background] Wisco, R., & Haber, C. (n.d.). A feasibility study of an emotion focused-mindfulness group. In Press.
- [Result] Vasiliadis HM, Dionne PA, Preville M, Gentil L, Berbiche D, Latimer E. The excess healthcare costs associated with depression and anxiety in elderly living in the community. Am J Geriatr Psychiatry. 2013 Jun;21(6):536-48. doi: 10.1016/j.jagp.2012.12.016. Epub 2013 Feb 6. PMID 23567409
- [Result] Troyer AK, Rich JB. Psychometric properties of a new metamemory questionnaire for older adults. J Gerontol B Psychol Sci Soc Sci. 2002 Jan;57(1):P19-27. doi: 10.1093/geronb/57.1.p19. PMID 11773220
- [Result] Pachana NA, Byrne GJ, Siddle H, Koloski N, Harley E, Arnold E. Development and validation of the Geriatric Anxiety Inventory. Int Psychogeriatr. 2007 Feb;19(1):103-14. doi: 10.1017/S1041610206003504. PMID 16805925
- [Result] Carpenter JS, Andrykowski MA. Psychometric evaluation of the Pittsburgh Sleep Quality Index. J Psychosom Res. 1998 Jul;45(1):5-13. doi: 10.1016/s0022-3999(97)00298-5. PMID 9720850
- [Derived] Hatch S, Finlayson M, Rej S, Kessler D. Virtually-Delivered Emotion Focused Mindfulness Therapy (EFMT) Group vs. Wait-List Control for Late-Life Anxiety: A Randomized Controlled Trial. Am J Geriatr Psychiatry. 2023 Oct;31(10):767-782. doi: 10.1016/j.jagp.2023.04.007. Epub 2023 Apr 19. PMID 37169708
- [Derived] Hatch S, Kessler D, Finlayson M, Rej S. Video-delivered emotion-focused mindfulness therapy for late- life anxiety: study protocol for a feasibility randomized controlled trial. Pilot Feasibility Stud. 2021 Sep 3;7(1):169. doi: 10.1186/s40814-021-00905-0. PMID 34479632